CLINICAL TRIAL: NCT05955547
Title: Comparison of the New Score (APACHE-INf), Including Inflammatory and Nutritional Parameters, With APACHE-II in the Prognosis of Patients Admitted to ICU
Brief Title: The New ICU Prognostic Score APACHE-INf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Nermin Kelebek Girgin (Unknown); Ayşegül Özkan (Unknown); Gülbahar Çalışkan (Unknown)
Responsible Party: Principal Investigator, Nizameddin Koca, MD, Associate Professor, Bursa City Hospital
Other Study IDs: APACHE-INf
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Intensive Care Unit; Inflammation; Nutritional Deficiency
Keywords: APACHE-INf; Prognosis scoring; Intensive Care Unit; inflammation; nutrition
MeSH Terms: conditions — Inflammation; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APACHE-II
  Interventions: Other: Prognosis Scoring
- APACHE-Inf
  Interventions: Other: Prognosis Scoring

INTERVENTIONS:
Other: Prognosis Scoring — To determine the prognosis of patients admitted to ICU with a scoring system that includes inflammation and nutritional status

SUMMARY:
Intensive care units (ICUs) aim to provide specialized care for patients with high morbidity and mortality risks. To effectively identify patients requiring urgent diagnosis and treatment, various scoring systems have been developed, including APACHE-II. However, these systems primarily focus on evaluating organ dysfunction and do not consider the patient's nutritional status or the role of inflammation. Recent studies have highlighted the crucial role of inflammation in patient outcomes, emphasizing the need to incorporate inflammatory parameters into scoring systems for accurate prognosis prediction. Additionally, nutritional status upon ICU admission has been largely overlooked in current scoring systems, despite its significant impact on patient outcomes. Malnourished patients have higher risks of complications, prolonged hospital stays, and increased mortality rates. Adequate nutrition supports immune function, tissue repair, and the response to therapeutic interventions, ultimately minimizing complications. Integrating nutritional assessment into existing scoring systems allows for early identification of malnourished patients and timely interventions, improving overall care quality in the ICU. Considering the importance of inflammation and nutritional status, this study aims to develop a new scoring system by adding inflammatory and nutritional parameters to APACHE II score. This comprehensive approach holds promise for enhancing patient outcomes, accurately evaluating clinical severity, and facilitating immediate interventions in critical care settings.

DETAILED DESCRIPTION:
Intensive care units are units where patients with high morbidity and mortality risk are followed up and treated. Risk stratification of patients in intensive care admission is very important in terms of quickly identifying patients who will require urgent diagnosis and treatment. For this reason, many scoring systems have been developed in recent years, and although the most common APACHE-II score is routinely applied in our intensive care units, there is no universally accepted consensus yet. Existing scoring systems predict prognosis mostly by evaluating organ dysfunction. The importance of inflammation and inflammatory response in organ functions has been better understood, especially in the COVID process. Nutritional status upon admission has not been evaluated in the current scoring systems.

Inflammation plays an important role in both regeneration and the fight against microorganisms at the cellular and tissue level. Recent studies have clearly demonstrated the importance of inflammation and inflammatory response in the morbidity and mortality of patients. In this context, there are studies reporting that some prominent inflammatory parameters are associated with morbidity and mortality rates in intensive care patients.

Based on the available evidence, it is evaluated that a scoring system that does not include inflammatory parameters cannot provide an accurate prognosis prediction.

the evaluation of nutritional status upon ICU admission is a vital component of patient care that has been largely overlooked in current scoring systems.

Malnourished patients are at a higher risk of developing complications, prolonged hospital stays, and increased mortality rates compared to well-nourished patients. Adequate nutrition not only supports immune function and tissue repair but also impacts the patient's response to therapeutic interventions and the prevention of complications during their ICU stay. Recognizing the significance of adequate nutrition in critical illness is essential to optimize patient outcomes and minimize complications. By integrating nutritional assessment into existing scoring systems, healthcare providers can identify malnourished patients early, implement timely interventions, and improve the overall quality of care in the ICU. This comprehensive approach holds promise for enhancing patient outcomes, reducing morbidity and mortality rates, and optimizing resource utilization in critical care settings.

Incorporating inflammation and nutritional status evaluation into existing scoring systems can provide a more comprehensive assessment of a patient's overall condition. Therefore, in this study, we aimed to evaluate whether a new scoring system, which will be created by adding inflammatory and nutritional parameters to APACHE II and SOFA scores, will provide a more accurate prognosis prediction.The electronic files of the patients who were followed up in Bursa City Hospital Intensive Care Units between 01.01.2020-31.12.2022 will be scanned retrospectively. Demographic data, clinical and laboratory data detailed below will be recorded in the files. After determining the cut-off points and scoring scale for each of the inflammatory tests at the time of admission obtained from the patient files, the competencies of the new and old scores obtained in prognosis prediction will be compared. By determining the cut-off points for the new scoring, it will be possible to evaluate the clinical severity of the patients more accurately and to carry out the necessary procedures immediately.

Data to be scanned from files:

Demographic data of the patient: Age, height, weight, Glasgow Coma score, APACHE 2 score, SOFA score, Concomitant diseases, Respiratory rate, Fever, Heart rate, SBP, DBP, OABP, Blood gas data: pH, pO2, PCO2, Osmolarity, Lactate, HCO3 Laboratory data: Detailed Hemogram data (WBC, Hgb, Hct, MCV, MPV, RDW, Plt, neutrophil, lymphocyte), Glucose, BUN, Cre, AST, ALT, T.bil, D.bil, Na, K, Ca, Mg, T. Protein, Albumin, Prealbumin, INR, aPTT, Vitamin D, Total cholesterol, LDL, HDL and Triglyseride Inflammation Parameters: Sedimentation, CRP, ferritin, D-dimer, fibrinogen, IL-6, procalcitonin

ELIGIBILITY:
Inclusion Criteria:

* ICU admission
* Age over 18

Exclusion Criteria:

* Incomplete data
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were admitted to ICU between 2019 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality Prediction | data of the ICU patients from 2019 to 2023 were evaluated
  Development with a score system that includes inflammation and nutritional status data in addition to APACHE-II scores would give a chance to evaluate ICU patient's overall status and predict the mortality risk more accurately

CONTACTS AND LOCATIONS:
Overall Officials: Nizameddin Koca, MD, Principal Investigator — University of Health Sciences, Bursa Sehir Training & Research Hospital
Locations (1):
- University of Health Sciences, Bursa Sehir Training & Research Hospital, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study would be performed as a multicenter study after single center data evaluation. IPD data would be shared with the participants of multicenter design researchers after the completion of single center study.